CLINICAL TRIAL: NCT02209207
Title: Continuous Versus Interval Walking Training in Patients With Severe Chronic Obstructive Pulmonary Disease - a Pilot Study
Brief Title: Continuous Versus Interval Walking Training in Patients With COPD - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physican (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Walking trial 2014
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: chronic obstructive pulmonary disease; endurance training; interval training; continuous training; walking training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous walking training (Active Comparator): n=10 patients with COPD Walking intensity 60 percent of 6-minute walking test speed
  Interventions: Device: Treadmill; Other: walking training
- Interval walking training (Active Comparator): n=10 patients with COPD Walking intensity 120 percent of 6-minute walking test speed for 1 minute alternating with 1 minute of rest
  Interventions: Device: Treadmill; Other: walking training

INTERVENTIONS:
Device: Treadmill
Other: walking training

SUMMARY:
This study will investigate the effects of interval walking training versus continuous walking training in patients with chronic obstructive pulmonary disease. Patients will be recruited during a 3-week inpatient pulmonary rehabilitation program and will be randomized to one of the two intervention groups. All walking training sessions will be performed on the same treadmill. Walking intensity in the continuous walking group will be 60 percent of the average speed of the 6-minute walking test. Patients in the interval training group will perform high intensity intervals at 120% of the 6-minute walking test speed for 60 seconds alternating with 60 seconds of rest. The total exercise duration will be progressively increased from 10 to 32 minutes.

ELIGIBILITY:
Inclusion Criteria:

* COPD stage III or IV according to the Global Initiative for chronic obstructive lung disease [GOLD]
* stationary patient in the Schön Klinik Berchtesgadener Land

Exclusion Criteria:

* acute, severe exacerbation of COPD
* failure to comply with study process

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
perceived exertion for dyspnea during walking training | day 1 to 21
  measured via modified Borg scale (0 to 10)

SECONDARY OUTCOMES:
heart rate during walking training | day 1 to 21
perceived exertion for leg fatigue (Borg-scale) | during three weeks of rehabilitation
Oxygen saturation during walking training | day 1 to 21
  measured via pulse oximeter
fat free mass in kilogram | day 1 to 21
  measured via Bioimpedance Analysis
forced expiratory volume in 1 second (FEV1) in liter | day 1 to 21
  measured by spirometry
Sit-to-stand-test | day 1 to 21
  5 repetitions of standing up and sitting down from a chair with crossed arms as quick as possible
6-minute walking test | day 1 to 21
  the best 6-minute walking test out of two tests on admission and at discharge will be taken
36 item short-form health Survey (SF-36) | day 1 to 21
  questionnaire for disease unspecific quality of life
chronic respiratory questionnaire (CRQ) | day 1 to 21
  disease specific quality of life questionnaire
hospital anxiety and depression scale (HADS) | day 1 to 21
  questionnaire on symptoms of anxiety and depression

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany